CLINICAL TRIAL: NCT02523339
Title: Multicenter Study of Retinal Oxygenation in Central Retinal Vein Occlusion
Brief Title: Study of Retinal Oxygenation in Central Retinal Vein Occlusion
Status: Completed | Type: Observational
Sponsor: University of Iceland (Other)
Collaborators: University Hospital, Basel, Switzerland (Other); Aston University (Other); University of Jena (Other); Medical University of Vienna (Other); University of Aarhus (Other); Clinical Research Center Memorial A. de Rothschild (Unknown); Palacky University (Other); University of Toyama (Other)
Responsible Party: Principal Investigator, Sveinn Hakon Hardarson, Post-doctoral researcher, University of Iceland
Other Study IDs: UI-CRVO-2015
Record Dates: First submitted 2015-08-07; First posted 2015-08-14 (Estimated); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Retinal Vein Occlusion
MeSH Terms: conditions — Retinal Vein Occlusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The purpose of the study is to test if oxygen saturation in retinal vessels is correlated with clinical parameters, such as visual acuity, central retinal thickness and presence of neovascularization. Retinal oximetry is performed with fundus camera based oximeters. The study will not entail change in treatment of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Suspected central retinal vein occlusion.
* Informed consent for participation.
* No treatment before the first oximetry measurement.

Exclusion Criteria:

* History of other retinal disease. Glaucoma and diabetes without retinopathy are not exclusion criteria but should be registered.
* History of cardiovascular or respiratory diseases that can be expected to influence systemic or retinal oxygen saturation. Examples: Known COPD or carotid stenosis. Subjects with high blood pressure will not be excluded but blood pressure should be registered.
* Poor quality images will be excluded based on the images themselves. Therefore, grading of cataract or other media opacities is not strictly necessary for the purpose of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected central retinal vein occlusion (CRVO) will be invited to participate.
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2014-10; Primary Completion 2018-06 (Actual); Study Completion 2020-11-03 (Actual)

PRIMARY OUTCOMES:
Retinal vessel oxygen saturation | 12 months
Visual acuity | 12 months
Central retinal thickness | 12 months
Presence or absence of ocular neovascularisation | 12 months
  As determined by gonioscopic examination

SECONDARY OUTCOMES:
Retinal vessel oxygen saturation | Baseline
Visual acuity | Baseline
Central retinal thickness | Baseline
Presence or absence of ocular neovascularisation | Baseline
  As determined by gonioscopic examination
Retinal vessel oxygen saturation | 3 months
Visual acuity | 3 months
Central retinal thickness | 3 months
Presence or absence of ocular neovascularisation | 3 months
  As determined by gonioscopic examination
Retinal vessel oxygen saturation | 6 months
Visual acuity | 6 months
Central retinal thickness | 6 months
Presence or absence of ocular neovascularisation | 6 months
  As determined by gonioscopic examination

CONTACTS AND LOCATIONS:
Overall Officials: Sveinn H. Hardarson, PhD, Principal Investigator — University of Iceland
Locations (8):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria
- Department of Ophthalmology, University Hospital and Faculty of Medicine and Dentistry, Palacky University Olomouc, Olomouc, Czechia
- Aarhus University. Department of Clinical Medicine - The Department of Ophthalmology, Aarhus, Denmark
- University Hospital Jena, Jena, Germany
- University of Iceland / Landspitali, Dept. of Ophthalmology, Reykjavik, Iceland
- Switzerland (2):
  - Eye Clinic of the University Hospital Basel, Basel, Canton of Basel-City
  - Clinical Research Center Memorial A. de Rothschild, Geneva
- Aston University School of Life and Health Sciences, Birmingham, United Kingdom